CLINICAL TRIAL: NCT03539809
Title: Determining the Optimal Ratio of Branched Chain Amino Acids in Medical Foods for Methylmalonic and Propionic Acidemias (MMA/PROP)
Brief Title: Branched Chain Amino Acids Ratio in Medical Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H18-00439
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Children
Keywords: Branched Chain Amino Acids; Direct Amino Acid Oxidation; Stable isotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCAA Ratio (Experimental): Different Branched-chain amino acid (BCAA) ratios will be tested. BCAA are comprised of 3 different amino acids (leucine, isoleucine and valine). The ratios among these 3 amino acids will be tested at 6 different ratios. Each intervention will be for 8hours.
  Interventions: Dietary Supplement: L-Amino Acids

INTERVENTIONS:
Dietary Supplement: L-Amino Acids — 6 different ratios of the Branched-chain Amino Acids (BCAA) will be tested for 8 hours each.

SUMMARY:
This study will evaluate the branched-chain amino acids (BCAA) ratio in the medical foods formulated for Methylmalonic and Propionic Acidemias (MMA/PROP) patients. We will recruit 6 healthy children between 6-10y (3 boys and 3 girls). They will be given amino acid-based shakes and protein free cookies. Using a minimally invasive stable isotope based technique, we will be able to determine the optimal ratio of BCAA to be added in the medical foods for the MMA/PROP subjects.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to use the minimally invasive Indicator Amino Acid Oxidation (IAAO) method in healthy school-aged children to determine the optimal ratio of BCAA in current medical foods used by MMA/PROP subjects. We will recruit healthy children to test our hypothesis.

Hypothesis:

1. The IAAO will be high (suggesting low protein synthesis) at high leucine levels and will be low (suggesting optimal protein synthesis) when leucine levels are reduced and at a better-balanced ratio of leucine to isoleucine and valine.
2. Children will have low levels of urine excretion of isoleucine and valine, with high leucine urinary excretion, when given the high ratio of leucine to valine and isoleucine. With the reduction of leucine intake in the diet, the urinary concentration of both isoleucine and valine will normalize.

Justification:

The use of medical foods as a sole source of energy and protein in patients with MMA/PROP has been discouraged. The recommendations state that such medical foods should be only used for patients who can't consume their RDA from natural protein. Since most of these patients are poor eaters, and at risk for malnutrition, they depend on medical foods as an easy tolerable source of energy and protein. The medical foods formulated for MMA/PROP contain imbalanced BCAA ratio (high leucine to minimal or no valine and isoleucine). The high leucine levels antagonize the other two BCAA and even suppresses their plasma and urine levels below normal. Determining the optimal ratio of BCAA is necessary to optimize protein synthesis, growth and prevent the accumulation of toxic metabolites. This proposal will focus on applying stable isotope tracers in healthy children to examine different intakes of leucine while keeping the amount of valine and isoleucine restricted as per the recommendations. Using the minimally invasive indicator amino acid technique (IAAO), and L-1-13C-Phenylalanine as the indicator amino acid for protein synthesis, the optimal amount of leucine to be added in one of the most commonly used medical food for these patients will be tested. In addition, the leucine intake which normalizes urine isoleucine and valine excretion will also be determined to be useful for patient management. Starting with the studies on healthy children ages 6-10 years to allow for characterization of the metabolic response to the different leucine intakes. Consequently, based on the results we obtain, we will be able to design the studies in MMA/PROP patients with the appropriate BCAA ratios to test.

Objectives:

1. Our primary objective is to examine the impact of reducing leucine levels from the current high doses in medical foods, sequentially, while holding isoleucine and valine at MMA/PROP recommended intakes, on protein synthesis using the IAAO technique in healthy children (6-10y).
2. Our secondary objective is to determine the impact of reducing leucine levels from the current high doses in medical foods, sequentially, while holding isoleucine and valine at MMA/PROP recommended intakes, on urinary excretion of BCAA.

Research Design:

This is a repeated measure study design involving 1 pre-study visit and 6 studies visits for each child, approximately one week apart from each other.

Statistical Analysis:

Results will be expressed as means ± SDs. Repeated Measures ANOVA will be used to assess the relationship of phenylalanine oxidation, and BCAA urinary excretion to the variable BCAA intakes using SAS statistical software (version 9.4; SAS Institute, Cary, NC). In all cases, the difference will be considered significant at P < 0.05. Repeated measure ANOVA will be used to measure the difference between means of F13CO2 oxidations in response to 6 leucine test intakes, as well as means of BCAA urinary excretions. When warranted, post hoc analysis will be performed using Tukey's multiple comparisons test to confirm where the differences occur between different conditions (leucine test intakes).

ELIGIBILITY:
Inclusion Criteria:

* Healthy school-aged children 6-10y
* Normal weight
* Normal eating habits
* English speaking children

Exclusion Criteria:

* Children under 6 years old, or over 10 years old.
* Children who are currently ill, with a fever, cold, vomiting or diarrhea.
* Children outside of normal weight parameters (3rd -85th percentiles for weight).
* Children with claustrophobia.
* Children currently or recently taking medication or antibiotics.
* Children with food allergies.
* Children who cannot speak, write and read in English

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
13C Phenylalanine Oxidation | 8 hours
  Breath and Urine samples will be collected during the study to measure 13C Phenylalanine oxidation

SECONDARY OUTCOMES:
Urinary Branched Chain amino acids excretion | 8 hours
  Urine samples will be collected during the study to measure BCAA urinary excretion

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No